CLINICAL TRIAL: NCT04964401
Title: The Effect of Ultrasound Guided Erector Spinae Plane Block Versus Thoracic Paravertebral Block on Acute and Chronic Pain After Video-Assisted Thoracic Surgery
Brief Title: US-Guided ESPB Versus TPVB on Acute and Chronic Pain After VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-KAEK-15:2232
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain; Video-Assisted Thoracoscopic Surgery; Thoracic Paravertebral Block; Erector Spinae Plane Block; Acute Pain; Chronic Pain
Keywords: Chronic pain; Erector spinae plane block; Thoracic paravertebral block; Acute pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Paravertebral Block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the thoracic 5 spinous process, the US-compatible needle will be advanced to the paravertebral area with in-plane technique, and 20 ml of 0.25% bupivacaine hydrochloride will be injected into this area.
  Interventions: Procedure: Thoracic paravertebral block vs Erector spinae plane block
- Erector spinae plane block (Active Comparator): After the linear ultrasound (US) probe will be placed 2-3 cm lateral to the T5 spinous process, 20 ml of 0.25% bupivacaine hydrochloride will be injected into the interfacial space below the erector spinae muscle, above the transverse process.
  Interventions: Procedure: Thoracic paravertebral block vs Erector spinae plane block

INTERVENTIONS:
Procedure: Thoracic paravertebral block vs Erector spinae plane block — Thoracic paravertebral block and erector spinae plane block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, when the patient is placed in the lateral decubitus position.

SUMMARY:
Postoperative acute and chronic pain is frequently observed in patients undergoing video assisted thoracoscopic surgery (VATS). This prolongs the discharge time of patients and increases the frequency of postoperative pulmonary complications. Recently, alternative analgesic methods such as thoracic paravertebral block (TPVB) and erector spinae plane block (ESPB), which are thought to have less side effects than thoracic epidural analgesia, have been used. Among these methods, ultrasound (US) guided TPVB is the most preferred method. In addition, ESPB application is increasing in patients undergoing VATS. In the literature, the number of cases performed with ESPB and randomized controlled prospective studies with ESPB are increasing. In this study, it is planned to compare the effects of US-guided TPVB and ESPB on postoperative acute and chronic pain in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-30 kg/m2
* Patients undergoing elective video assiste thoracoscopic surgery

Exclusion Criteria:

* Advanced cancer
* History of chronic analgesic therapy
* History of local anesthetic allergy
* Infection in the intervention area
* Patients with bleeding disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Pain scores | 24 hours after surgery
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 1st, 2nd, 4th, 8th, 16th and 24th hours after surgery.

SECONDARY OUTCOMES:
Chronic pain | First and 3th month
  Chronic pain findings will be evaluated in the 1st month and 3rd month after surgery by using visual analog from 0 (no pain) to 10 (worst pain). Neuropathic pain symptoms (Burning, stabbing, or electric shock-like pain; tingling, numbness, or a "pins and needles" feeling, hyperalgesia, allodynia and hypoesthesia) will also be asked to the participants in the 1st month and 3rd month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No